CLINICAL TRIAL: NCT01563510
Title: Comparison of Laparoscopic Versus Open Operation for Hepatolithiasis
Brief Title: Research of the Key Technology and Standardization of Minimal Invasive Treatment for Hepatolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shuguo Zheng, MD (Other)
Responsible Party: Sponsor-Investigator, Shuguo Zheng, MD, Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department;, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWHZSG001; zhengshuguo (Registry Identifier: zhengshuguo)
Record Dates: First submitted 2012-03-21; First posted 2012-03-27 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Biliary Stones
Keywords: Hepatolithiasis; Minimal invasive surgery; Laparoscopic hepatectomy; Choledochoscope
MeSH Terms: conditions — Cholecystolithiasis | interventions — Heller Myotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic operation (Experimental): Total laparoscopic anatomical hepatectomy were performed, combined with cholecystectomy and bile duct exploration when necessary. The intraoperative ultrasound, choledochoscope and hepatic segmental staining were used selectively.
  Interventions: Procedure: Laparoscopic operation
- Open operation (Active Comparator): The traditional open regular hepatectomy were performed, combined with cholecystectomy and bile duct exploration when necessary. The intraoperative ultrasound and choledochoscope were used selectively.
  Interventions: Procedure: Open operation

INTERVENTIONS:
Procedure: Laparoscopic operation — Fifty patients with early regional hepatolithiasis were selected and divided into laparoscopic hepatectomy group as described in the detailed description. Total laparoscopic anatomical hepatectomy were performed, combined with cholecystectomy and bile duct exploration when necessary. The intraoperative ultrasound, choledochoscope and hepatic segmental staining were used selectively.
  Other Names: Laparoscopic hepatectomy for early regional hepatolithiasis
  Arms: Laparoscopic operation
Procedure: Open operation — Fifty patients with early regional hepatolithiasis were selected and divided into open group as described in the detailed description. The traditional open regular hepatectomy were performed, combined with cholecystectomy and bile duct exploration when necessary. The intraoperative ultrasound and choledochoscope were used selectively.
  Other Names: Open operation for regional hepatolithiasis
  Arms: Open operation

SUMMARY:
The purpose of this research is to investigate the key technology and the related issues of minimal invasive treatment for hepatolithiasis and to build new methods of minimal invasive operation for hepatolithiasis. The validity, feasibility and limitations of the laparoscopic operation were assessed objectively through our clinical prospective study. The technique points, indications and contraindications were summarized to evaluate the status and role of minimal invasive laparoscopic operation in the treatment of hepatolithiasis.

DETAILED DESCRIPTION:
Background: China is the high incidence area of hepatolithiasis. The development of minimal invasive techniques opened up a new situation for the treatment of hepatolithiasis, but it has not been widely applied.

Intervention: Comparison of minimal invasive versus open operation for hepatolithiasis: a prospective randomized study. One hundred patients with early regional hepatolithiasis were selected and divided into laparoscopic operation group and open operation group randomly, each group contains 50 cases. Laparoscopic anatomical hepatectomy or open regular hepatectomy were performed respectively, combined with cholecystectomy and bile duct exploration when necessary. The intraoperative ultrasound and choledochoscope were used selectively.

Results:

1. Clinical data: previous operation history, operation time, intraoperative blood loss, volume of blood transfusion, complications and mortality, postoperative liver function, residual stones, recurrence rate, long-term curative effect and survival time were collected and analysed.
2. Statistical method: univariate/multivariate analysis, logistic regression analysis, mixed linear regression, Cox survival analysis were used.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with regional stones distributed in a segment, lobe or half liver, combined or not combined with extrahepatic biliary calculi, hepatic parenchymal atrophy or fibrosis in the lesion region
2. Liver function > Child-pugh level B, no severe biliary cirrhosis, ICG ≤ 15%, the residual liver volume and standard liver volume ratio ≥ 40%
3. Patients with good general condition, the conditions of open Anatomical Hepatectomy were achieved
4. Other organ lesions and previous biliary tract operation is not the absolute exclusion criteria
5. Written informed consent

Exclusion Criteria:

1. Age: older than 70 years old, younger than 18 years old
2. Patients with bad general condition or important organ lesions, liver resection could not be tolerated
3. Complicated case needed to get emergency operation
4. Combined with severe liver atrophy hypertrophy syndrome, hepatic portal transposition or hilar biliary fibrosis / stenosis
5. Combined with severe biliary cirrhosis and portal hypertension, severe varicose of hepatic portal vein , hepatic insufficiency
6. Diagnosed with cholangiocellular carcinoma intraoperatively or by postoperative pathology
7. Contraindication of laparoscopy: Combined with complicated acute cholangitis, repeated biliary tract operation, heavy intra-abdominal adhesion, Trocar can not be placed in. Artificial pneumoperitoneum could not be tolerated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with residual stones or cholangitis symptoms | up to 5 years postoperation
  Liver function, recurrence rate, cholangitis symptoms, quality of life and survival time were collected and analysed to evaluate the postoperative curative effect. The follow up interval time: every six months.

SECONDARY OUTCOMES:
Number of participants with operation complication | Duration hospitalization(an expected average of 2 weeks) to 2 months postoperation
  Operation time, intraoperative blood loss, volume of blood transfusion, complications and mortality, postoperative liver function, residual stones were collected and analysed to evaluate the safety and effectiveness of the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, MD, Study Director — Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Uchiyama K, Kawai M, Ueno M, Ozawa S, Tani M, Yamaue H. Reducing residual and recurrent stones by hepatectomy for hepatolithiasis. J Gastrointest Surg. 2007 May;11(5):626-30. doi: 10.1007/s11605-006-0024-8. PMID 17468921
- [Background] Lee SK, Seo DW, Myung SJ, Park ET, Lim BC, Kim HJ, Yoo KS, Park HJ, Joo YH, Kim MH, Min YI. Percutaneous transhepatic cholangioscopic treatment for hepatolithiasis: an evaluation of long-term results and risk factors for recurrence. Gastrointest Endosc. 2001 Mar;53(3):318-23. doi: 10.1016/s0016-5107(01)70405-1. PMID 11231390
- [Background] Uenishi T, Hamba H, Takemura S, Oba K, Ogawa M, Yamamoto T, Tanaka S, Kubo S. Outcomes of hepatic resection for hepatolithiasis. Am J Surg. 2009 Aug;198(2):199-202. doi: 10.1016/j.amjsurg.2008.08.020. Epub 2009 Feb 27. PMID 19249730
- [Background] Otani K, Shimizu S, Chijiiwa K, Ogawa T, Morisaki T, Sugitani A, Yamaguchi K, Tanaka M. Comparison of treatments for hepatolithiasis: hepatic resection versus cholangioscopic lithotomy. J Am Coll Surg. 1999 Aug;189(2):177-82. doi: 10.1016/s1072-7515(99)00109-x. PMID 10437840
- [Background] Buell JF, Cherqui D, Geller DA, O'Rourke N, Iannitti D, Dagher I, Koffron AJ, Thomas M, Gayet B, Han HS, Wakabayashi G, Belli G, Kaneko H, Ker CG, Scatton O, Laurent A, Abdalla EK, Chaudhury P, Dutson E, Gamblin C, D'Angelica M, Nagorney D, Testa G, Labow D, Manas D, Poon RT, Nelson H, Martin R, Clary B, Pinson WC, Martinie J, Vauthey JN, Goldstein R, Roayaie S, Barlet D, Espat J, Abecassis M, Rees M, Fong Y, McMasters KM, Broelsch C, Busuttil R, Belghiti J, Strasberg S, Chari RS; World Consensus Conference on Laparoscopic Surgery. The international position on laparoscopic liver surgery: The Louisville Statement, 2008. Ann Surg. 2009 Nov;250(5):825-30. doi: 10.1097/sla.0b013e3181b3b2d8. PMID 19916210
- [Background] Lai EC, Ngai TC, Yang GP, Li MK. Laparoscopic approach of surgical treatment for primary hepatolithiasis: a cohort study. Am J Surg. 2010 May;199(5):716-21. doi: 10.1016/j.amjsurg.2009.02.007. Epub 2009 Dec 3. PMID 19959158
- [Background] Cho JY, Han HS, Yoon YS, Shin SH. Experiences of laparoscopic liver resection including lesions in the posterosuperior segments of the liver. Surg Endosc. 2008 Nov;22(11):2344-9. doi: 10.1007/s00464-008-9966-0. Epub 2008 Jun 5. PMID 18528623
- [Background] Zhang L, Chen YJ, Shang CZ, Zhang HW, Huang ZJ. Total laparoscopic liver resection in 78 patients. World J Gastroenterol. 2009 Dec 7;15(45):5727-31. doi: 10.3748/wjg.15.5727. PMID 19960572
- [Background] Nguyen KT, Gamblin TC, Geller DA. World review of laparoscopic liver resection-2,804 patients. Ann Surg. 2009 Nov;250(5):831-41. doi: 10.1097/SLA.0b013e3181b0c4df. PMID 19801936